CLINICAL TRIAL: NCT04440098
Title: Isolated During COVID-19: Effects of COVID-19's Social Restrictions on Loneliness and Psychosocial Symptomatology
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Viviana Horigian, Professor, Educator Track, University of Miami
Other Study IDs: 20200446
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Loneliness; Depression; Anxiety; Alcohol Abuse; Drug Abuse
MeSH Terms: conditions — Depression; Anxiety Disorders; Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Isolated Observational group: All participants socially restricted as a result of COVID-19

SUMMARY:
This study seeks to gather data and insight on epidemiologic trends of loneliness and other behaviors in the wake of the CDC recommended "social distancing" during the COVID-19 pandemic. The objective of this study is to use a cross-sectional survey to assess the impact of COVID-19's associated recommendations (social distancing, self-isolation, and self-quarantine) on loneliness and psychosocial symptomatology (depression, anxiety, substance abuse) on young adults (18-35 years old).

ELIGIBILITY:
Inclusion Criteria

* 18-35 years old
* Currently living in the United States

Exclusion Criteria

* Those under 18 years, or older than 35 years
* Adults unable to consent
* Non-English-speaking adults

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 1008 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Loneliness as evaluated by the UCLA loneliness scale | Day 1
  University of California Los Angeles ( UCLA) Loneliness Scale is a 20-item self-report questionnaire that evaluates subjective feelings of loneliness and social isolation. Participants rate items on a 4-point Likert scale ranging from 1 (never) to 4 (often).Items are summed to create a score that can range from 20-80, higher scores being indicative of greater loneliness.
Alcohol Use as evaluated by the AUDIT | Day 1
  Alcohol Use Disorder Identification Test (AUDIT) is a 10-item self-reported questionnaire used to identify individuals whose alcohol consumption could be hazardous for their health. Participants rate items in a 5-point Likert scale, indicating amount (0 to 10 drinks or more), frequency (never to daily or almost daily), and indication of problems caused by alcohol (yes or no). Items were summed up to create a score that can range from 0 to 50. A score of 1 to 7 indicates low risk consumption, whereas a score of 8-15 suggests risky or hazardous drinking, a score of more than 15 is likely to indicate high-risk drinking and alcohol dependence.
Drug Use as evaluated by the DAST-10 | Day 1
  The Drug Abuse Screening Test (DAST-10) is a 10-item self-reported screening test that provides a quantitative index of the degree of consequences related to drug abuse. Participants rate items yes or no, positive responses corresponding to 1 point. Items are summed up to create a score that can range from 0-10. A score of 1-2 represents risky behaviors related to drugs, 3-5 represents moderate problems, 6-8 represents substantial problems, and 9-10 represents severe problems.
Anxiety as evaluated by GAD-7 | Day 1
  The General Anxiety Disorder Scale (GAD- 7) is a 7- item self-reported screening tool that assess presence and severity of Generalized Anxiety Disorder. Participants rated frequency of problems in a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). Items are summed up to create a score with scores of 5, 10, and 15 being the cut-off points for mild, moderate and severe anxiety, respectively.
Depression as assessed by CES-D-10 | Day 1
  The Center for Epidemiologic Studies Depression scale (CES-D-10) is a 10-item self-reported measure that assesses the frequency of symptoms of depression. Participants rate frequency of symptoms in a 4-point Likert scale from 0 (rare or none of the time) to 3 (most or almost all the time). Items are summed up to create a score that ranges from 0 to 30, with higher scores representing greater depressive symptoms. A score of 16 or more represents clinical depression.

CONTACTS AND LOCATIONS:
Overall Officials: Viviana E Horigian, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horigian VE, Schmidt RD, Feaster DJ. Loneliness, Mental Health, and Substance Use among US Young Adults during COVID-19. J Psychoactive Drugs. 2021 Jan-Mar;53(1):1-9. doi: 10.1080/02791072.2020.1836435. Epub 2020 Oct 28. PMID 33111650